CLINICAL TRIAL: NCT00962546
Title: Computed Tomographic Perfusion and Computed Tomographic Angiography as Screening Tools for Vasospasm Following Subarachnoid Hemorrhage
Brief Title: Computed Tomographic (CT) Perfusion and CT Angiography as Screening Tools for Vasospasm Following Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Michelle Miller-Thomas, MD, Assistant Professor, Washington University School of Medicine
Other Study IDs: HRPO 09-0950
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Cerebral Vasospasm; Cerebral Aneurysm; Subarachnoid Hemorrhage
Keywords: cerebral aneurysm; subarachnoid hemorrhage; cerebral vasospasm; computed tomographic perfusion; computed tomographic angiography
MeSH Terms: conditions — Vasospasm, Intracranial; Intracranial Aneurysm; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CTA/CTP: Patients undergo CTA/CTP imaging prior to cerebral angiography

SUMMARY:
Cerebral vasospasm is a devastating complication of subarachnoid hemorrhage after cerebral aneurysm rupture leading to cerebral ischemia and potentially cerebral infarction. The current gold standard diagnostic imaging study for cerebral vasospasm is catheter cerebral angiography, an invasive diagnostic procedure carrying a complication rate of 1-2% per procedure. Computed tomographic perfusion imaging (CTP) and computed tomographic angiography (CTA) are noninvasive diagnostic imaging studies frequently utilized in the evaluation of embolic and thrombotic cerebral infarct. The investigators hypothesize that CTP and CTA may be utilized as screening tools for cerebral vasospasm following aneurysmal subarachnoid hemorrhage requiring treatment and provide prognostic information.

ELIGIBILITY:
Inclusion Criteria:

* subarachnoid hemorrhage after aneurysm rupture

Exclusion Criteria:

* renal insufficiency
* pregnancy
* contrast reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the neurological intensive care unit with subarachnoid hemorrhage due to rupture of a cerebral aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
CT perfusion parameters | at time of catheter angiogram

SECONDARY OUTCOMES:
Disposition at discharge | At time of hospital discharge
vessel narrowing by CT angiography | at time of catheter angiogram

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Miller-Thomas, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Result] Wintermark M, Ko NU, Smith WS, Liu S, Higashida RT, Dillon WP. Vasospasm after subarachnoid hemorrhage: utility of perfusion CT and CT angiography on diagnosis and management. AJNR Am J Neuroradiol. 2006 Jan;27(1):26-34. PMID 16418351
- [Result] Aralasmak A, Akyuz M, Ozkaynak C, Sindel T, Tuncer R. CT angiography and perfusion imaging in patients with subarachnoid hemorrhage: correlation of vasospasm to perfusion abnormality. Neuroradiology. 2009 Feb;51(2):85-93. doi: 10.1007/s00234-008-0466-7. Epub 2008 Oct 11. PMID 18850093
- [Result] Mustonen T, Koivisto T, Vanninen R, Hanninen T, Vapalahti M, Hernesniemi J, Kuikka JT, Vanninen E. Heterogeneity of cerebral perfusion 1 week after haemorrhage is an independent predictor of clinical outcome in patients with aneurysmal subarachnoid haemorrhage. J Neurol Neurosurg Psychiatry. 2008 Oct;79(10):1128-33. doi: 10.1136/jnnp.2007.142851. Epub 2008 Mar 20. PMID 18356250